CLINICAL TRIAL: NCT07249892
Title: A Multicenter, Open-label Phase I/II Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, Dosimetry and Efficacy of BPR-6023021 in Subjects With Advanced Solid Tumors With Bone Metastases.
Brief Title: A Study of BPR-6023021 in Advanced Solid Tumors With Bone Metastases
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chengdu Syncor Pharmaceutical Co., Ltd. (Industry)
Collaborators: Beijing Quarkxia Technology Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BPR-6023021-101; CTR20254494 (Registry Identifier: National Medical Products Administration (NMPA) Drug Clinical Trial Registration And Information Publicity Platform)
Record Dates: First submitted 2025-11-14; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Solid Tumors
Keywords: BPR-6023021; Advanced Solid Tumors; Bone Metastases
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1:Dose escalation (Experimental): 5 dose levels of BPR-6023021 are tentatively planned for Phase 1
  Interventions: Drug: BPR-6023021 for injection
- Phase 2: RP2D Cohort (Experimental): Participants will receive BPR-6023021 for injection at the Recommended Phase 2 Dose (RP2D) determined from the Phase 1 dose escalation study.The dose of BPR-6023021 for injection in Phase 2 is selected based on the Phase 1 monotherapy dose escalation study.
  Interventions: Drug: BPR-6023021 for injection

INTERVENTIONS:
Drug: BPR-6023021 for injection — BPR-6023021 is a Radionuclide conjugated drugs (RDC) targeting bone.

SUMMARY:
A multicenter, open-label Phase I clinical trial to evaluate the safety, tolerability, pharmacokinetics, dosimetry and efficacy of BPR-6023021 in subjects with advanced solid tumors with bone metastases

DETAILED DESCRIPTION:
This study is a multicenter, open-label Phase I clinical trial to evaluate the safety, tolerability, pharmacokinetics, dosimetry and efficacy of BPR-6023021 in subjects with advanced solid tumors with bone metastases. The study is divided into two parts: Phase I and Phase II. The Phase I study is the dose escalation phase. The primary objective is to assess the safety and tolerability of a single administration of BPR-6023021 and to determine the Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD) based on the occurrence of Dose-Limiting Toxicities (DLTs) associated with BPR-6023021 (if the MTD cannot be determined).The Phase II study is the dose expansion phase. The primary objective is to explore the efficacy of BPR-6023021 at a selected dose level.

ELIGIBILITY:
Inclusion Criteria

1. The age should be up to 18 years at the time of signing the informed consent form (ICF);
2. The Eastern Cooperative Oncology Group (ECOG) performance status score should be ≤ 1;
3. The expected survival period should be ≥ 3 months
4. Phase I and phase II: Subjects with advanced solid tumor bone metastases diagnosed by histology or cytology; and the subjects have failed standard treatment, or have no standard treatment, or are intolerant or not applicable to standard treatment
5. Before the first administration, a 99mTc-MDP bone scan diagnosed multiple bone metastases, and at least two site was confirmed by CT or MRI;
6. Have adequate organ and bone marrow functions;
7. For subjects with reproductive capacity, take effective medical contraceptive measures during the study treatment and within 6 months after the last administration;
8. The subjects voluntarily join this study, sign the informed consent form, and can comply with the visit and related procedures stipulated in the protocol.

Exclusion Criteria

1. The washout period before the first administration of the study drug was insufficient.
2. Previous received similar radionuclide internal irradiation treatment.
3. Previous received or planned to receive during the study period semi-body external radiotherapy targeting bone metastases.
4. Known "super bone imaging".
5. Known spinal cord compression, or clinical imaging manifestations suggesting impending spinal cord compression.
6. Any cardiovascular or cerebrovascular diseases or cardiovascular risk factors that may affect the treatment of the study drug.
7. Poorly controlled diabetes and hypertension.
8. The toxicity of previous anti-tumor treatment before the first administration has not recovered to ≤ 1 grade (evaluated based on NCI-CTCAE v5.0) or has not reached the level specified in the inclusion/exclusion criteria.
9. Had other malignant tumors within 5 years before the first administration.
10. Subjects with severe and/or uncontrolled concomitant diseases.
11. Active hepatitis B or active hepatitis C.
12. Human immunodeficiency virus (HIV) test positive or having a history of acquired immune deficiency syndrome (AIDS); known active syphilis infection.
13. During the screening process before the first administration, the condition deteriorated rapidly, such as significant changes in the investigator's assessment of physical condition, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 195 (Estimated)
Dates: Start 2025-11-19 (Estimated); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-09-06 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | Up to 1 year

SECONDARY OUTCOMES:
Dosimetry，including Maximum plasma concentration (Cmax) of BPR-6023021 | Through study completion, an average of 2 year
  To collect the biological distribution of major tissues/organs and so on.
Time to Radiographic Bone Progresion (TTRBP) | Through study completion, an average of 2 year
  Time from start of treatment to progression of bone lesion (PD) or death, whichever occurs first, during the study period
Radiographic progression-free survival (rPFS) | Through study completion, an average of 2 year
  Time from start of treatment to progression of Disease (PD) or death, whichever occurs first
Symptomatic skeletal event-free survival (SSE-FS) | Through study completion, an average of 2 year
  Time from start of treatment to the first occurrence of new SSE or death from any cause , whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Yang, Study Director — Chengdu Syncor Pharmaceutical Co., Ltd.; Wei Fan, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) collected in this study are considered confidential commercial information of the sponsor. Therefore, they will not be shared publicly to protect intellectual property and maintain competitive advantage.